CLINICAL TRIAL: NCT03027947
Title: Spinal Root and Spinal Cord Stimulation for Restoration of Function in Lower-Limb Amputees
Acronym: SCS-LL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Lee Fisher, PhD, Assistant Professor, School of Medicine, Physical Medicine and Rehabilitation, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19030223; UH3NS100541 (NIH)
Record Dates: First submitted 2016-10-05; First posted 2017-01-23 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Traumatic Amputation of Lower Extremity; Phantom Limb Pain
Keywords: Phantom Limb Pain; Lower-Limb Amputation; Electrodes; Stimulation; Pain; Sensation
MeSH Terms: conditions — Phantom Limb; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal cord stimulation (Experimental): Spinal cord stimulator leads (2-3 leads) will be placed in the lumbar epidural space of lower limb amputees to determine if the patient experiences any pain reduction from spinal cord stimulation.
  Participants in this study receive spinal cord stimulation will be trans-tibial and trans-femoral amputees that are at least six month post--amputation. Subjects will have varying levels of phantom limb sensation and pain, but should have no other significant neurological disorders.
  Interventions: Device: Spinal cord stimulator

INTERVENTIONS:
Device: Spinal cord stimulator — Spinal cord stimulator leads (2-3 leads) will be placed in the lumbar epidural space of lower limb amputees to determine if the patient experiences any pain reduction from spinal cord stimulation.

SUMMARY:
The goals of this study are to provide sensory information to amputees and reduce phantom limb pain via electrical stimulation of the lumbar spinal cord and spinal nerves. The spinal nerves convey sensory information from peripheral nerves to higher order centers in the brain. These structures still remain intact after amputation and electrical stimulation of the dorsal spinal nerves in individuals with intact limbs and amputees has been demonstrated to generate paresthetic sensory percepts referred to portions of the distal limb. Further, there is recent evidence that careful modulation of stimulation parameters can convert paresthetic sensations to more naturalistic ones when stimulating peripheral nerves in amputees. However, it is currently unclear whether it is possible to achieve this same conversion when stimulating the spinal nerves, and if those naturalistic sensations can have positive effects on phantom limb pain. As a first step towards those goals, in this study, the investigators will quantify the sensations generated by electrical stimulation of the spinal nerves, study the relationship between stimulation parameters and the quality of those sensations, measure changes in control of a prosthesis with sensory stimulation, and quantify the effects of that stimulation on the perception of the phantom limb and any associated pain.

DETAILED DESCRIPTION:
During the study, FDA-cleared spinal cord stimulator leads will be placed in the lumbar epidural space of lower limb amputees and steered laterally towards the dorsal spinal roots under fluoroscopic guidance. This approach is essentially identical to the FDA-cleared procedure in which these devices are placed in the lumbar epidural space for treatment of intractable low back and leg pain. In that procedure, it is common clinical practice to place 2-3 leads temporarily in the epidural space through a percutaneous approach and perform a multiday trial to determine if the patient experiences any pain reduction from spinal cord stimulation. Following the trial, the percutaneous leads are typically removed by gently pulling on them, and the patient is referred to a neurosurgeon for permanent surgical implantation.

Similarly, in this study, the device will be tunneled percutaneously through the skin and secured in place with tape or suture. Using the stylet included with the spinal cord stimulator leads, the devices will be steered laterally under fluoroscopic guidance to target the dorsal spinal nerves. During lab experiments, the leads will be connected to an external stimulator. In this study, the devices will remain in the epidural space for less than 30 days and will be removed by gently pulling on the external portion. Throughout the study, the investigators will perform a series of psychophysical evaluations to characterize the sensory percepts evoked by epidural stimulation, along with functional evaluations of the effects of stimulation on the ability to control a prosthetic limb. In addition, the investigators will perform surveys to characterize changes in phantom limb sensation and pain that occur during stimulation.

ELIGIBILITY:
Inclusion Criteria:

* have an amputation of at least one lower limb, at a level between the ankle and hip joints
* be at least 6 months post-amputation at time of lead placement

Exclusion Criteria:

* women who are pregnant or breast-feeding
* has any serious diseases or disorders that affect ability to participate
* currently receiving medications that may affect blood coagulation
* allergic to contrast medium, or has kidney failure that could be exacerbated by contrast agent
* implanted metallic devices that are not cleared for MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Stimulation perceptual thresholds to a variety of stimulus parameters | 30 days
  Quantify the threshold (minimum charge and pulse rate) stimulus required to evoke sensory percepts during epidural spinal nerve stimulation.
Stimulation neurophysiology thresholds to a variety of stimulus parameters | 30 days
  Quantify the threshold (minimum charge and pulse rate) stimulus required to evoke neurophysiological responses during epidural spinal nerve stimulation

SECONDARY OUTCOMES:
Location of evoked sensory percepts | 30 days
  Document where on the body the subject perceives the stimulation locations.
Qualitative self-report of evoked sensations | 30 days
  Document the subjective perception of lumbosacral epidural spinal nerve stimulation for restoration of sensation. The investigators will ask each subject to provide subjective feedback on their perceived utility of the sensory feedback provided by the device.
Change (reduction) in pain ratings | 30 days
  Document changes in phantom limb pain during and shortly after lumbosacral epidural spinal nerve stimulation in amputees. Before placement of the spinal cord stimulator leads, investigators will document the subject's description of their history of perceived phantom limb. Investigators will ask them to periodically update their perception of the limb throughout each experimental session, as well as within a month after the device has been removed.
Ability to use a prosthetic limb with neural signals | 30 days
  Investigators will test the subject's success rate during control of prosthetic limb with and without sensory feedback provided by electrical stimulation of the spinal roots. Using either a virtual prosthetic limb or an instrumented prosthesis, stimulation of the spinal roots will be modulated based on signals recorded from the limb.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Fisher, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Debbie, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team may share de-identified data with scientists at other centers for the purpose of data analysis and collaboration. Research information and data may be shared with investigators conducting other research.
Supporting Information: Study Protocol, ICF
Time Frame: Information may be shared while data is being recorded, analyzed, and/or prior to publication. Data may be available after manuscripts are published.
Access Criteria: Data may be shared through a restricted access portal created by the National Institutes of Health or directly with scientists at other centers under a data use agreement.

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Etter K, Borgia M, Resnik L. Prescription and repair rates of prosthetic limbs in the VA healthcare system: implications for national prosthetic parity. Disabil Rehabil Assist Technol. 2015 Nov;10(6):493-500. doi: 10.3109/17483107.2014.921246. Epub 2014 May 22. PMID 24852068
- [Background] Raichle KA, Hanley MA, Molton I, Kadel NJ, Campbell K, Phelps E, Ehde D, Smith DG. Prosthesis use in persons with lower- and upper-limb amputation. J Rehabil Res Dev. 2008;45(7):961-72. doi: 10.1682/jrrd.2007.09.0151. PMID 19165686
- [Background] Deer TR, Grigsby E, Weiner RL, Wilcosky B, Kramer JM. A prospective study of dorsal root ganglion stimulation for the relief of chronic pain. Neuromodulation. 2013 Jan-Feb;16(1):67-71; discussion 71-2. doi: 10.1111/ner.12013. Epub 2012 Dec 14. PMID 23240657
- [Background] Liem L, Russo M, Huygen FJ, Van Buyten JP, Smet I, Verrills P, Cousins M, Brooker C, Levy R, Deer T, Kramer J. A multicenter, prospective trial to assess the safety and performance of the spinal modulation dorsal root ganglion neurostimulator system in the treatment of chronic pain. Neuromodulation. 2013 Sep-Oct;16(5):471-82; discussion 482. doi: 10.1111/ner.12072. Epub 2013 May 13. PMID 23668228